CLINICAL TRIAL: NCT02249819
Title: Evaluating Anodal tDCS Preceding Aphasia Therapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Bruce Volpe, Principal Investigator, Northwell Health
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-416
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2019-02

CONDITIONS: Stroke; Aphasia
Keywords: stroke; aphasia; CVA; apraxia; cerebrovascular accident; cerebral stroke; speech therapy; aphasia therapy; non-invasive brain stimulation; transcranial direct current stimulation; tDCS
MeSH Terms: conditions — Stroke; Aphasia; Apraxias; Communication Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: All participants received both stimulation conditions (active tDCS + computerized naming therapy and sham tDCS + computerized naming therapy), separated by a 1-week washout period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sequence of stimulation conditions was randomized across subjects.
Oversight: Data Monitoring Committee: No

ARMS (2):
- anodal tDCS, then sham tDCS (Experimental): Participants received 1 single 20 min session of anodal tDCS + computerized naming therapy. Following a 1 week washout period, they received 1 single 20 min session of sham tDCS + computerized aphasia therapy. Sequence of stimulation conditions was randomized across participants.
  Interventions: Device: transcranial direct current stimulation
- sham tDCS, then anodal tDCS (Experimental): Participants received 1 single 20 min session of sham tDCS + computerized naming therapy. Following a 1 week washout period, they received 1 single 20 min session of anodal tDCS + computerized aphasia therapy. Sequence of stimulation conditions was randomized across participants.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Soterix 1x1 anodal tDCS

SUMMARY:
The purpose of this study is to determine if non-invasive brain stimulation (transcranial direct current stimulation) delivered prior to language therapy will improve word-finding in individuals with aphasia who are 6 months or greater post-stroke.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. First single focal unilateral left hemisphere lesion with diagnosis verified by brain imaging (MRI or CT scans) that occurred at least 6 months prior
3. Pre-morbidly right handed
4. Pre-morbidly fluent English speaker
5. Cognitive function sufficient to understand the experiments and follow instructions (per interview with Speech Pathologist)
6. A baseline Aphasia Quotient score between 10 to 94 out of 100 points on the Western Aphasia Battery (neither completely without language comprehension/expression nor fully recovered from aphasia).

Exclusion Criteria:

1. Ongoing use of CNS-active medications
2. Ongoing use of psychoactive medications, such as stimulants, antidepressants, and anti-psychotic medications
3. Presence of additional potential tDCS risk factors:

   * Damaged skin at the site of stimulation (i.e., skin with ingrown hairs, acne, razor nicks, wounds that have not healed, recent scar tissue, broken skin, etc.)
   * Presence of an electrically, magnetically or mechanically activated implant (including cardiac pacemaker), an intracerebral vascular clip, or any other electrically sensitive support system
   * Metal in any part of the body, including metal injury to the eye (jewelry must be removed during stimulation)
   * A history of medication-resistant epilepsy in the family
   * Past history of seizures or unexplained spells of loss of consciousness during the previous 36 months
4. Pregnancy in women, as determined by self-report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Feinstein Institute for Medical Research, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Monti A, Cogiamanian F, Marceglia S, Ferrucci R, Mameli F, Mrakic-Sposta S, Vergari M, Zago S, Priori A. Improved naming after transcranial direct current stimulation in aphasia. J Neurol Neurosurg Psychiatry. 2008 Apr;79(4):451-3. doi: 10.1136/jnnp.2007.135277. Epub 2007 Dec 20. PMID 18096677
- [Background] Baker JM, Rorden C, Fridriksson J. Using transcranial direct-current stimulation to treat stroke patients with aphasia. Stroke. 2010 Jun;41(6):1229-36. doi: 10.1161/STROKEAHA.109.576785. Epub 2010 Apr 15. PMID 20395612
- [Background] Fiori V, Coccia M, Marinelli CV, Vecchi V, Bonifazi S, Ceravolo MG, Provinciali L, Tomaiuolo F, Marangolo P. Transcranial direct current stimulation improves word retrieval in healthy and nonfluent aphasic subjects. J Cogn Neurosci. 2011 Sep;23(9):2309-23. doi: 10.1162/jocn.2010.21579. Epub 2010 Oct 14. PMID 20946060
- [Background] Holland R, Crinion J. Can tDCS enhance treatment of aphasia after stroke? Aphasiology. 2012 Sep;26(9):1169-1191. doi: 10.1080/02687038.2011.616925. Epub 2011 Nov 3. PMID 23060684
- [Background] Marangolo P, Fiori V, Campana S, Calpagnano MA, Razzano C, Caltagirone C, Marini A. Something to talk about: enhancement of linguistic cohesion through tdCS in chronic non fluent aphasia. Neuropsychologia. 2014 Jan;53:246-56. doi: 10.1016/j.neuropsychologia.2013.12.003. Epub 2013 Dec 11. PMID 24333381

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants received both the active and sham tDCS conditions, and sequence of stimulation conditions was randomized across participants.
Groups:
- Anodal tDCS, Then Sham tDCS: Participants first received 1 single 20 min session of anodal tDCS + computerized naming therapy. After a washout period of 1 week, they then received 1 single 20 min session of sham tDCS + computerized naming therapy.
- Sham tDCS, Then Anodal tDCS: Participants first received 1 single 20 min session of sham tDCS + computerized naming therapy. After a washout period of 1 week, they then received 1 single 20 min session of anodal tDCS + computerized naming therapy.
Period: Overall Study
Arm/Group | Anodal tDCS, Then Sham tDCS | Sham tDCS, Then Anodal tDCS
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Crossover design study: All participants were randomized to receive one single 20 min session of anodal tDCS and 1 single session of sham tDCS followed by computerized naming therapy. Sequence of stimulation conditions was counterbalanced across participants with a 1 week washout period in between conditions.
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Picture-naming Accuracy Score
Description: The mean change in verbal picture-naming accuracy score (out of 75) was calculated from baseline to discharge in each condition (sham and active tDCS).
Time Frame: baseline, discharge
Population: All participants received one dose of each intervention and completed all study visits. They were consequently all included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: score
Groups:
- Anodal tDCS: Participants received 1 single 20 min session of anodal tDCS + computerized naming therapy in either the first two or the last two weeks of the study.
- Sham tDCS: Participants received 1 single 20 min session of sham tDCS + computerized naming therapy in either the first two or the last two weeks of the study.
Arm/Group | Anodal tDCS | Sham tDCS
Number analyzed (Participants) | 15 | 15
score
  Mean Score at Discharge(out of 75) | 51.33 (17.79) | 51.00 (18.40)
  Mean Change from Baseline | 5.25 (4.85) | 5.92 (5.21)
Statistical Analysis 1: Comparison: Anodal tDCS vs Sham tDCS; Test type: Equivalence — Statistical analysis for mean change from baseline in naming accuracy in the anodal vs. sham tDCS conditions Null hypothesis is that there was no difference in mean change of naming accuracy between anodal and sham tDCS conditions. A significance level of 0.05 was used (two-sided); p = 0.694, wilcoxon sign-ranked test — The wilcoxon sign-ranked test was performed for this crossover design study in which subjects underwent measures across 2 study conditions (paired samples: mean change in anodal vs. sham condition). A significance level of 0.05 was used (two-sided); Western Aphasia Battery used as a screening tool on admission only, to characterize level of severity. It was NOT an outcome measure

ADVERSE EVENTS:
Time Frame: Two weeks for each intervention
Description: Safety population included all participants who received at least one dose of intervention.
Groups:
- Anodal tDCS: Participants who received anodal tDCS + computerized picture-naming therapy, and were followed for 2 weeks.
- Sham tDCS: Participants who received sham tDCS + computerized picture-naming therapy, and were followed for 2 weeks.
Arm/Group | Anodal tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-07-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT02249819/Prot_SAP_000.pdf
  • Informed Consent Form (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT02249819/ICF_001.pdf